CLINICAL TRIAL: NCT03432611
Title: Evaluation of a Smartphone Application for Self Care for Women With Menstrual Pain (Primary Dysmenorrhea): a Randomized Trial
Brief Title: A Smartphone App for Women With Primary Dysmenorrhea
Acronym: smartAID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: smartAID-18
Record Dates: First submitted 2018-01-18; First posted 2018-02-14 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Primary Dysmenorrhea
Keywords: mHealth; dysmenorrhea; acupressure; self-management; self-care
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: randomized, three-armed pragmatic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complete app (Experimental): 198 women with primary dysmenorrhea who receive an app which includes a self-care information feature and a self-acupressure feature.
  Interventions: Other: Self-care information feature; Other: Self-acupressure feature
- Control intervention I (Active Comparator): 198 women with primary dysmenorrhea who receive an app for menstrual pain which includes the self-care information feature, but not the self-acupressure feature.
  Interventions: Other: Self-care information feature
- Control intervention II (Active Comparator): 198 women with primary dysmenorrhea who receive an app for menstrual pain which includes the self-acupressure feature, but not the self-care information feature.
  Interventions: Other: Self-acupressure feature

INTERVENTIONS:
Other: Self-care information feature — The self-care feature offers information on self-care for menstrual pain. The following topics are shown: exercise, dietary supplementation, heating pad/hot water bottle, yoga, and information on when to consult a doctor and how primary dysmenorrhoea is often treated. Notifications from the app which can be deactivated remind women of surveys and activities.
  Arms: Complete app; Control intervention I
Other: Self-acupressure feature — The acupressure feature offers detailed written and multimedia descriptions of an acupressure used for menstrual pain. Three acupressure points are described, which should be massaged bilaterally twice a day up to five times a day on the 5 days before menstruation and during menstruation. Each point should be massaged for 2 minutes. A timer for the acupressure and notifications from the app which can be deactivated remind women of surveys and acupressure.
  Arms: Complete app; Control intervention II

SUMMARY:
With a randomized, pragmatic study the effectiveness of a smartphone app for menstrual pain in 18-34-year-old women with primary dysmenorrhea will be investigated.

DETAILED DESCRIPTION:
Smartphone apps may be useful to guide and support individuals in self-management strategies. Primary dysmenorrhea is a very common problem for women. With a randomized, pragmatic study the investigators aim to evaluate whether a smartphone app for women with menstrual pain is effective in reducing menstrual pain in 18-34-year-old women with primary dysmenorrhea. For this the investigators compare the complete smartphone app with two control versions of this app. The complete app provides evidence-based self-care information and instructions for self-acupressure in menstrual pain, the control intervention I includes self-care information, but no instructions for self-acupressure, and control intervention II includes instructions for self-acupressure, but no self-care information. The investigators aim to observe 594 women with primary dysmenorrhea over 12 menstruation cycles. The primary outcome is the mean pain intensity on the days with pain during the 6th menstruation after randomization using a numerical rating scale (NRS; 0=no pain; 10=strongest pain imaginable). Women are eligible when they suffer from primary dysmenorrhea, are between 18 and 34 years old, not pregnant and do not plan to be pregnant within the next 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-34 years
* Dysmenorrhea, defined as self-reported menstrual cramps or pain during every menstrual cycle which started during the teenage years
* No prior history of a gynecological disease that is known to be a reason for the dysmenorrhea
* Not more than 5 days with menstrual pain outside the menstrual period itself
* Menstruation within the last six weeks and a cycle length of 3 to 6 weeks
* Moderate or severe pain, defined as a score equal to or higher than 6 on a numeric rating scale (NRS, 0 to 10) for the worst pain intensity during the last menstruation
* Informed consent
* Possession of an iPhone
* Willingness and ability to input and share anonymous data through the study app
* The willingness to see a doctor when 1) pain is getting worse than usual, 2) pain medication is not helping, and 3) when the pain is still present well before or well after the period.

Exclusion Criteria:

* Known pregnancy
* Pregnancy already planned for the forthcoming 12 months

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with menstrual pain
Enrollment: 594 (Estimated)
Dates: Start 2018-02-19 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Mean pain intensity on the days with pain | Daily during the 6th menstruation after randomization
  The mean pain intensity on the days with pain during the 6th menstruation after randomization using a numerical rating scale (NRS; 0=no pain; 10=strongest pain imaginable).

SECONDARY OUTCOMES:
Mean pain intensity on the days with pain | Baseline; daily during menstruation (1st to 5th and 7th to 12th menstrual cycles)
  The mean pain intensity on the days with pain during the menstruation 1 to 5 and 7 to 12 after randomization using a numerical rating scale (NRS; 0=no pain; 10=strongest pain imaginable).
Responder | Daily during menstruation (1st to 12th menstrual cycles)
  Responder defined as having at least 50% pain reduction on the days with pain
Number of days with pain (duration of pain) | Daily during menstruation (1st to 12th menstrual cycles)
  Number of days participants reported pain.
Days with absence from work, training, or studies | Baseline, end of menstruation (1st to 12th menstrual cycles)
  Days with absence from work or education because of menstrual pain during previous period.
Days with pain medication | Daily during menstruation (1st to 12th menstrual cycles)
  Days with intake of pain medication for menstrual pain during each menstruation
Adverse reaction | End of menstruation (1st to 12th menstrual cycles)
  Characteristics of adverse reaction
Severe adverse events | End of menstruation (3rd, 6th, 9th, and 12th menstrual cycles)
  Characteristics and duration of severe adverse events
Frequency of acupressure application | 5 days before menstruation and during menstruation (1st to 12th menstrual cycles)
  Number of times acupressure was applied during each cycle
User satisfaction | End of menstruation (1st to 12th menstrual cycles)
  User's satisfaction with app guided activity (NRS; 0=totally unsatisfied; 6=very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M. Witt, MD, Principal Investigator — Charite University, Berlin, Germany; Daniel Pach, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang J, Rogge AA, Armour M, Smith CA, D'Adamo CR, Pischke CR, Yen HR, Wu MY, More AOO, Witt CM, Pach D. International ResearchKit App for Women with Menstrual Pain: Development, Access, and Engagement. JMIR Mhealth Uhealth. 2020 Feb 11;8(2):e14661. doi: 10.2196/14661. PMID 32058976